CLINICAL TRIAL: NCT02702440
Title: Effect of Liquid Versus Solid Calories on Body Weight: a Systematic Review and Meta-analysis of Controlled Feeding Trials
Brief Title: Meta-analyses of Liquid Versus Solid Calories and Body Weight
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: John Sievenpiper (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, John Sievenpiper, Associate Professor, University of Toronto
Organization: University of Toronto (Other)
Other Study IDs: CIHR-Liquid Calories 2015
Record Dates: First submitted 2016-03-02; First posted 2016-03-08 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes Mellitus; Chronic Disease; Cardiovascular Diseases; Prediabetic State; Overweight; Obesity; Metabolic Syndrome
Keywords: Systematic review and meta-analysis; Sugars; Liquid calories; Solid calories; Clinical trials; Body weight; Body Mass Index; Evidence-base nutrition (EBN); Evidence-base medicine (EBM); Clinical practice guidelines
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease; Cardiovascular Diseases; Prediabetic State; Overweight; Obesity; Metabolic Syndrome; Body Weight

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Liquid calories from sugars

SUMMARY:
Consumption of sugar-sweetened beverages (SSBs) has been linked to rising rates of overweight and obesity. The most prominent mechanism to explain the link between SSBs and obesity is that liquid calories are not perceived by the body; thereby, promoting less satiety, less energy compensation and more weight gain than does the same energy consumed in solid form. This view is supported by pooled analyses of acute preload trials that have primarily measured food intake as the outcome. Though failure of short-term compensation has been observed with liquid calories, results from these acute preload trials should not be extrapolated to infer that liquid energy sources lead to weight gain over the long-term. To date, it is unclear whether liquid calories have differential effects than solid calories on body weight gain over the longer term. To increase clarity in this issue, the investigators propose to conduct a systematic review and meta-analysis from long-term controlled feeding trials to distinguish the contribution of liquid calories from solid calories on body weight over the long-term. The findings generated by this analysis will improve the health of consumers through informing evidence-based guidelines and improving health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

DETAILED DESCRIPTION:
Background: The prevalence of overweight and obese individuals has dramatically risen over the past 30 years and represents a major threat to public health. Sugars consumed in liquid form (i.e. SSBs) have been targeted as a prominent contributor towards obesity. Pooled analyses of acute preload trials that have assessed food intake as the primary outcome suggest that liquid calories from sugars are more poorly compensated than solid calories. Though tempting, results from these acute studies should not be extrapolated to infer that liquid energy sources lead to weight gain over the long term. A study of long-term randomized controlled trials by Kaiser et al. found that when adults were required to consume sugar sweetened beverages (SSBs) as an additional source of energy, dose-dependent weight gain was observed. However, this weight gain was far less than half the amount one would have predicted to be gained using a mathematical model. This suggests that over extended periods of time, majority of the energy consumed as SSBs is indeed compensated for.

Need for proposed research: To date, it is unknown whether people compensate differently for liquid versus solid sources of calories over the long term.

Objective: To synthesize evidence of the effect of liquid calories versus solid calories on body weight in controlled trials.

Design: This systematic review and meta-analysis will be conducted according to the Cochrane Handbook for Systematic Reviews of Interventions and reported according to the Preferred Reporting Items for Systematic Reviews and Meta-Analyses (PRISMA).

Data sources: MEDLINE, EMBASE, and The Cochrane Central Register of Controlled Trials (Clinical Trials; CENTRAL) will be searched using appropriate search terms supplemented by hand searches of references of included studies.

Study selection: The investigators will include controlled trials (randomized and non-randomized) that have compared the effects of liquid sources of calories in isocaloric exchange for solid sources of calories on body weight for >= 7 days in humans (healthy or non-healthy).

Data extraction: Following systematic exclusion based on title and abstract, 2 reviewers will independently review and extract relevant data from each report that meets the inclusion criteria. Risk of bias will be assessed using the Cochrane Risk of Bias Tool. All disagreements among reviewers were resolved by consensus. Missing variance data will be calculated using standard computations and imputations.

Outcomes: Body weight (kg)

Data synthesis: Pooled analyses of the mean difference will be performed using the generic inverse variance method. Random-effects models will be used even in the absence of statistically significant between-study heterogeneity because they yield more conservative summary effect estimates in the presence of residual heterogeneity. Fixed-effects models will be used only if there are less than 5 included trials. Crossover trials will be assessed via paired analyses. Heterogeneity will be assessed by the Cochran Q statistic and quantified by the I2 statistic. Sensitivity and subgroup analyses will be conducted to identify sources of heterogeneity. Sensitivity analyses will involve an assessment of heterogeneity upon systematic removal of each trial. If there are >= 10 trials, the study investigators will conduct apriori subgroup analyses by age, health status, comparator, dose, baseline measurements, randomization, study design (parallel, crossover), energy balance (positive, neutral, negative), follow-up (<= 4 weeks, > 4 weeks) and risk of bias. Meta-regression analyses will assess the significance of categorical and continuous subgroup analyses. When more than 10 trials are available, publication bias will be investigated by funnel plots and formal testing using Egger and Begg tests. If publication bias is suspected, then the investigators will attempt to adjust for funnel plot asymmetry by imputing the missing study data using the Duval and Tweedie trim and fill method.

Evidence assessment: The strength of the evidence for each outcome will be assessed using the Grading of Recommendations Assessment, Development and Evaluation (GRADE).

Knowledge translation plan: The results will be disseminated through interactive presentations at local, national, and international scientific meetings and publication in high impact factor journals. Target audiences will include the public health and scientific communities with interest in nutrition and obesity. Feedback will be incorporated and used to improve the public health message and key areas for future research will be defined. Applicant/Co-applicant Decision Makers will network among opinion leaders to increase awareness and participate directly as committee members in the development of future guidelines.

Significance: The proposed research will aid in distinguishing the role of liquid calories from solid calories on body weight over the long-term. This will strengthen the evidence-base for guidelines and improve health outcomes by educating healthcare providers and patients, stimulating industry innovation, and guiding future research design.

ELIGIBILITY:
Inclusion Criteria:

* Controlled trials in humans
* Treatment duration more or equal than 7 days
* Viable endpoint data (body weight)
* Suitable control (e,i. Isocaloric exchange of liquid carbohydrates with solid carbohydrates)

Exclusion Criteria:

* Non-human studies
* No viable endpoint data
* Acute preload studies (< 7 days)
* Lack of a suitable control (non-isocaloric)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All individuals, both children and adults, regardless of health status.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Body weight | Up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: John L Sievenpiper, MD, PhD, FRCPC, Principal Investigator — University of Toronto
Locations (1):
- The Toronto 3D (Diet, Digestive tract and Disease) Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Kaiser KA, Shikany JM, Keating KD, Allison DB. Will reducing sugar-sweetened beverage consumption reduce obesity? Evidence supporting conjecture is strong, but evidence when testing effect is weak. Obes Rev. 2013 Aug;14(8):620-33. doi: 10.1111/obr.12048. Epub 2013 Jun 7. PMID 23742715
- [Background] Almiron-Roig E, Palla L, Guest K, Ricchiuti C, Vint N, Jebb SA, Drewnowski A. Factors that determine energy compensation: a systematic review of preload studies. Nutr Rev. 2013 Jul;71(7):458-73. doi: 10.1111/nure.12048. Epub 2013 Jun 10. PMID 23815144
- [Background] Allison DB. Liquid calories, energy compensation and weight: what we know and what we still need to learn. Br J Nutr. 2014 Feb;111(3):384-6. doi: 10.1017/S0007114513003309. Epub 2013 Oct 29. No abstract available. PMID 24164833